CLINICAL TRIAL: NCT04771130
Title: A Phase 1b/2, Open-Label, Dose Finding, and Expansion Study of the Bcl-2 Inhibitor BGB-11417 in Patients With Myeloid Malignancies
Brief Title: A Study of BGB-11417 in Participants With Myeloid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-103; 2021-003285-12 (EudraCT Number); 2023-508881-14-00 (EU CTIS Number); CTR20213416 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm
Keywords: BGB-11417; Azacitidine; Posaconazole; AML; MDS; MDS/MPN
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases | interventions — Azacitidine; posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Parts 1 and 2: AML Cohorts (Experimental): Participants with AML will receive BGB-11417 and azacitidine on a 28-day cycle.
  Interventions: Drug: BGB-11417; Drug: Azacitidine
- Parts 1 and 2: MDS Cohorts (Experimental): Participants with MDS will receive BGB-11417 and azacitidine on a 28-day cycle.
  Interventions: Drug: Azacitidine; Drug: BGB-11417
- Part 3: AML and MDS Cohorts (Experimental): Participants with AML and MDS will receive BGB-11417 and azacitidine on a 28-day cycle. A subset of the participants will receive a modified second cycle of treatment to explore drug-drug interactions (DDI) with posaconazole.
  Interventions: Drug: BGB-11417; Drug: Azacitidine; Drug: Posaconazole
- Part 3: AML and MDS Cohort (Experimental): Participants with MDS and R/R AML (China only) will receive BGB-11417 on a 28-day cycle.
  Interventions: Drug: BGB-11417

INTERVENTIONS:
Drug: BGB-11417 — Oral administration for 10, 21, 14 or 28 days on a 28-day cycle.
  Other Names: Sonrotoclax
  Arms: Part 3: AML and MDS Cohorts; Parts 1 and 2: AML Cohorts
Drug: Azacitidine — Intravenous or subcutaneous administration for 7 days.
  Arms: Part 3: AML and MDS Cohorts; Parts 1 and 2: AML Cohorts; Parts 1 and 2: MDS Cohorts
Drug: Posaconazole — Oral administration for 8 days on second cycle only.
  Arms: Part 3: AML and MDS Cohorts
Drug: BGB-11417 — Oral administration for 28 days on a 28-day cycle.
  Arms: Part 3: AML and MDS Cohort
Drug: BGB-11417 — Oral administration for 10, 14 or 21 days on a 28-day
  Arms: Parts 1 and 2: MDS Cohorts

SUMMARY:
The study will determine the safety, tolerability, recommended Phase 2 dose (RP2D) and preliminary efficacy of BGB-11417 as monotherapy and in combination with azacitidine in participants with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS)or MDS/myeloproliferative neoplasm (MPN) .

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed diagnosis of one of the following by 2016 World Health Organization criteria:

   * AML, nonacute promyelocytic leukemia
   * MDS
   * MDS/MPN
2. Eastern Cooperative Oncology Group performance status of 0 to 2.
3. Adequate organ function defined as:

   * Creatinine clearance ≥ 50 milliliters/minute (mL/min) (or between 30 and 49 mL/min in unfit AML cohort)
   * Adequate liver function
4. Life expectancy of > 12 weeks.
5. Ability to comply with the requirements of the study.

Key Exclusion Criteria:

1. A diagnosis of acute promyelocytic leukemia.
2. History of prior malignancy, with the exception of either a history of MDS or MDS/MPN that has transformed to AML, or other prior malignancy that was treated with a full curative intent and no evidence of recurrence within the past 2 years (eg, localized skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score ≤ 6 prostate cancer)
3. Antecedent MPN including myelofibrosis, essential thrombocytosis, polycythemia vera, or chronic myelogenous leukemia with or without BCR-ABL1 translocation and AML with BCR-ABL1 translocation.
4. Prior therapy with a B-cell lymphoma-2 inhibitor
5. Known central nervous system involvement by leukemia.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2028-02-08 (Estimated); Study Completion 2028-02-08 (Estimated)

PRIMARY OUTCOMES:
Part 1 And 2: Number Of Participants Experiencing Dose-limiting Toxicities (DLTs) | Cycle 1 (Up to 28 days for non-hematologic DLTs and up to 42 days for hematologic DLTs)
Part 1 And 2: Number Of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Approximately 24 months
Part 3 AML Cohort: Complete Remission (CR) Plus CR With Partial Hematologic Recovery (CRh) Rate | Approximately 24 months
  CR plus CRh will be defined as the percentage of participants whose best overall response (BOR) is CR plus CRh. BOR will be defined as the best response recorded from the first dose of study drug until data cut or the initiation of new anticancer treatment.
Part 3 MDS Cohort: Modified Overall Response (mOR) Rate | Approximately 24 months
  The mOR will be defined as the percentage of participants whose BOR is achieving CR, marrow complete remission (mCR), or partial remission (PR) at any time point during the study for myelodysplastic/myeloproliferative neoplasm (MDS/MPN).
Part 3 AML Cohort (DDI Sub-cohort): Area Under Plasma Concentration-time Curve (AUC) from time 0 to the last quantifiable timepoint (t) (AUC0-t) Of BGB-11417 When Administered Alone and when Co-administered With Posaconazole | Cycle 2 Day 12 and Cycle 2 Day 20 (predose and 1, 2, 4, 6, 8, and 24 hours postdose)
Part 3 AML Cohort (DDI Sub-cohort): Maximum Observed Plasma Concentration (Cmax) Of BGB-11417 When Administered Alone and When Co-administered With Posaconazole | Cycle 2 Day 12 and Cycle 2 Day 20 (predose and 1, 2, 4, 6, 8, and 24 hours postdose)
Part 3 AML Cohort (DDI Sub-cohort): Area Under Plasma Concentration-time Curve (AUC) from time 0 to infinity (AUC0-infinity) Of BGB-11417 When Administered Alone and When Co-administered With Posaconazole | Cycle 2 Day 12 and Cycle 2 Day 20 (predose and 1, , 4, 6, 8, and 24 hours postdose)
Part 3 AML and MDS Cohorts (Treated with Monotherapy): Number Of Participants Experiencing DLTs | Cycle 2
Part 3 AML and MDS Cohorts (Treated with Monotherapy): Number of Participants Experiencing TEAEs | Approximately 24 months

SECONDARY OUTCOMES:
Parts 1 And 2 AML Cohort: Complete remission (CR) + Morphologic CR With Partial Hematologic Recovery (CRh) | Approximately 24 months
Parts 1 And 2 MDS Cohort: mOR Rate | Approximately 24 months
Parts 1 And 2: Cmax Of Azacitidine When Coadministered With BGB-11417 | Day 0 and 4 (Cycle 1) predose and at multiple time points up to 4 hours postdose
Parts 1 And 2: Terminal Half-life (t1/2) Of Azacitidine When Coadministered With BGB-11417 | Day 0 and 4 (Cycle 1) predose and at multiple time points up to 4 hours postdose
Parts 1 And 2: AUC From Time Zero To Time t (AUC0-t) Of Azacitidine When Coadministered With BGB-11417 | Day 0 and 4 (Cycle 1) predose and at multiple time points up to 4 hours postdose
Parts 1 And 2: AUC From Time Zero To Infinity (AUC0-inf) Of Azacitidine When Coadministered With BGB-11417 | Day 0 and 4 (Cycle 1) predose and at multiple time points up to 4 hours postdose
Parts 1 And 2: Apparent Total Clearance Of Azacitidine From Plasma (CL/F) When Coadministered With BGB-11417 | Day 0 and 4 (Cycle 1) predose and at multiple time points up to 4 hours postdose
Parts 1 And 2: Apparent Volume Of Distribution (Vz/F) Of Azacitidine When Coadministered With BGB-11417 | Day 0 and 4 (Cycle 1) predose and at multiple time points up to 4 hours postdose
Parts 1 And 2: Steady-state AUC From Time Zero To Time Of Last Measurable Concentration (AUClast,ss) Of BGB-11417 When Coadministered With Azacitidine | Day 1-4 and 28 (Cycle 1) Day 5 (Cycle 2) predose and at multiple time points up to 8 hours postdose
Parts 1 And 2: Steady-state Cmax (Cmax,ss) Of BGB-11417 When Coadministered With Azacitidine | Day 1-4 and 28 (Cycle 1) Day 5 (Cycle 2) predose and at multiple time points up to 8 hours postdose
Parts 1 And 2: Steady-state Trough Plasma Concentration (Ctrough,ss) Of BGB-11417 When Coadministered With Azacitidine | Day 1-4 and 28 (Cycle 1) Day 5 (Cycle 2) predose and at multiple time points up to 8 hours postdose
Parts 1 And 2: Steady-state Time To Maximum Observed Plasma Concentration (tmax,ss) Of BGB-11417 When Coadministered With Azacitidine | Day 1-4 and 28 (Cycle 1) Day 5 (Cycle 2) predose and at multiple time points up to 8 hours postdose
Part 3: Number Of Participants Experiencing TEAEs | Approximately 24 months
Part 3: Complete Response Rate | Approximately 24 months
  CR will be defined as the percentage of participants whose BOR is CR. BOR will be defined as the best response recorded from the first dose of study drug until data cut or the initiation of new anticancer treatment.
Part 3 AML Cohort: CR With Incomplete Hematologic Recovery (CRi) Rate | Approximately 24 months
  CRi will be defined as the percentage of participants whose BOR is CRi.
Part 3 AML Cohort: Overall Response Rate (ORR) | Approximately 24 months
  The ORR will include participants whose BOR include CR, CRi, PR, and morphologic leukemia-free state.
Part 3 AML Cohort: Duration Of Response (DOR) | Approximately 24 months
  DOR will be defined as the time from the first response to disease progression documented after treatment initiation or death, whichever occurs first. DOR will include CR, CR plus CRi, overall response (OR), and CR plus CRh.
Part 3 AML Cohort: Time To Response (TTR) | Approximately 24 months
  TTR will be defined as the time from treatment initiation to the first documented response and will include CR, CR plus CRi, OR, and CR plus CRh.
Part 3 Event-free Survival (EFS) | Approximately 24 months
  EFS will be defined as the time from treatment initiation to disease progression, treatment failure, relapse (hematologic relapse for AML) for those who have treatment success, or death due to any cause, whichever happens first.
Part 3 Overall Survival (OS) | Approximately 24 months
  OS will be defined as the time from treatment initiation to death. OS will be analyzed using the same methods as the EFS analysis except for the censoring rules.
Part 3 AML Cohort: Number of Participants with Transfusion Independence | Approximately 24 months
  Transfusion independence will be defined as the proportion of participants whose BOR is transfusion independence. Transfusion independence will need to last for at least 56 consecutive days postbaseline.
Part 3 MDS Cohort: Number Of Participants With Hematological Improvement-erythroid (HI-E) | Approximately 24 months
  The proportion of participants whose BOR is HI-E
Part 3 MDS Cohort: Proportion Of Participants With Hematological Improvement-platelet (HI-P) | Approximately 24 months
  The proportion of participants whose BOR is HI-P
Part 3 MDS Cohort: Proportion Of Participants With Hematological Improvement-neutrophil (HI-N) | Approximately 24 months
  The proportion of participants whose BOR is HI-N will be reported.
Part 3 MDS Cohort: Number of participants with Transfusion Independence | Approximately 24 months
  Transfusion independence will be defined as the percentage of participants whose BOR is transfusion independence. Transfusion independence will need to last for at least 56 consecutive days postbaseline.
Part 3: Ctrough,ss Of BGB-11417 When Coadministered With Azacitidine | Cycle 1 Day 1 and Cycle 2 Day 5 (predose and 4 and 6 hours postdose)
Part 3 MDS cohort: Partial Hematologic Recovery CRh | Approximately 24 months
  Percentage of participants with partial hematologic recovery will be reported
Part 3 AML (Treated with Monotherapy): Complete Response + Morphologic complete Remission with Partial Hematologic Recovery | Approximately 24 months
  Percentage of participants with Complete Response + Morphologic complete Remission with Partial Hematologic Recovery will be reported.
Part 3 AML (Treated with Monotherapy): Steady State trough plasma concentration of BGB-11417 | Cycle 2 Day 12 and Cycle 2 Day 20 (predose and 1, 4, 6, 8, and 24 hours postdose)
Part 3 MDS (Treated with Monotherapy): Modified Overall Response | Approximately 24 months
  Percentage of participants with modified overall response including CR, marrow CR (mCR) or partial remission (PR)
Part 3 MDS (Treated with Monotherapy): Steady State trough plasma concentration of BGB-11417 | Cycle 2 Day 12 and Cycle 2 Day 20 (predose and 1, 4, 6, 8, and 24 hours postdose)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Tampa General Hospital, Tampa, Florida
  - Upmc Hillman Cancer Center(Univ of Pittsburgh), Pittsburgh, Pennsylvania
  - Md Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (11):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Orange Health Hospital, Orange, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Linear Clinical Research, Nedlands, Western Australia
  - One Clinical Research, Nedlands, Western Australia
- China (12):
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Peoples Hospital of Shenzhen, Shenzhen, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- France (3):
  - Hopital Claude Huriez Chu Lille, Lille
  - Hopital Larchet, Nice
  - Hopital Saint Louis, Paris
- Germany (2):
  - Universitaetsklinikum Leipzig Aor, Leipzig
  - Universitaetsklinikum Ulm, Ulm
- Italy (3):
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Niguarda Cancer Center Division of Hematology, Milan
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Wellington Regional Hospital (Ccdhb), Wellington
- South Korea (2):
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
- Spain (4):
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari I Politecnic La Fe, Valencia
- United Kingdom (2):
  - Edinburgh Cancer Centre, Edinburgh
  - The Christie Hospital, Greater Manchester

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/